CLINICAL TRIAL: NCT06078137
Title: Impact of an Enhanced Patient Reported Outcome Measurement (PROM) Strategy on PROM Completion Rates, Decision Support, and Patient Experience: A Hybrid Effectiveness-Implementation Study
Brief Title: Impact of an Enhanced Patient Reported Outcome Measurement (PROM) Strategy on PROM Completion Rates
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, David Ring, Professor of Surgery and Perioperative Care Department, University of Texas at Austin
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: STUDY00001696
Record Dates: First submitted 2023-09-28; First posted 2023-10-11 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: PROM

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Patients randomized to intervention receive both usual Patient reported outcome measure (PROM) and new PROMs strategy (on the technology platform for English speakers and on REDCap/Qualtrix for Spanish Speakers) done after rooming.
  Interventions: Other: Usual PROMs and new PROMs strategy
- Control group (No Intervention): Patients go through the registration process which includes PROMs completion using Ipads. Enrolled in the room at the end of the visit.

INTERVENTIONS:
Other: Usual PROMs and new PROMs strategy — Patients randomized to intervention receive both usual PROMs and new PROMs strategy
  Arms: Intervention Group

SUMMARY:
in clinical practice has been curbed by issues related to the variability in use of these tools for decision-making, and universally poor completion rates over time. Patients may not see the relevance of responding to questions about their health, and the results may not be reviewed by the clinician or presented and visualized with the patient. The questions may seem impersonal (e.g. too general and not directly assessing their individual goals, motivations, aspirations), irrelevant (e.g., asking about symptoms of depression when a person is seeking musculoskeletal specialty care) and insensitive (e.g., asking about sensitive subjects at the outset thereby disengaging the individual), and redundant or awkward (e.g., presenting questions that seem very similar or administered in strange orders). Finally, PROMs may also confer some burden (e.g., long PROM questionnaires often used for research may be unnecessarily burdensome for patient care), and provide logistical challenges (e.g., difficulties in administering the tools at the right time points), adding to a poor patient experience.

DETAILED DESCRIPTION:
The investigator sought to assess the impact of an enhanced and more personalized PROM strategy to overcome these barriers by providing i) a primer ahead of PROMs administration, ii) simple 3-part survey capturing capability, comfort, and calm, iii) a short distress and misconception survey, iv) goal setting question, v) summary sheet of PRO scores, and vi) a commitment intervention. Patients will subsequently be requested to complete the CollaboRATE survey, JSPPE survey, and questions about their experience in relation to the new format of surveys (only if they were in the intervention group) before receiving a text message reminder around 6-weeks followed by a set of deprioritization questions and the 3-part capability, comfort, and calm survey.

ELIGIBILITY:
Inclusion Criteria:

All new patients English and Spanish speakers

Exclusion criteria:

Cognitive deficiency precluding PROM completion Language other than English or Spanish

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Completion of 3-survey patient-reported outcome measure at 6-week follow-up via Text | through study completion, an average of 6 weeks
  We will assess the completion of 3-survey patient-reported outcome measure at 6-week follow-up via Text.
Completion of answered text | through study completion, an average of 6 weeks
  We will assess the completion response rate.
Completion of deprioritization options 1 or 2 at 6-week follow-up via text or email | through study completion, an average of 6 weeks
  "1 = I got what I needed" "2 = I didn't receive anything useful" "3 = I'm still receiving care"
Jefferson Scale of Patient's Perceptions of Physician Empathy | through study completion, an average of 6 weeks
  The Jefferson Scale of Patient's Perceptions of Physician Empathy includes five 7-point scale questions and higher scores indicated greater perceived clinician empathy.

CONTACTS AND LOCATIONS:
Overall Officials: David Ring, MD, Principal Investigator — Professor of orthopedic surgery at The university of Texas at Austin
Locations (1):
- University of Texas Health Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No